CLINICAL TRIAL: NCT03999645
Title: Is it Safe to do Laparoscopic Cholecystectomy for Acute Cholecystitis up to Seven Days? A Randomized Clinical Trial
Brief Title: Is it Safe to do Laparoscopic Cholecystectomy for Acute Cholecystitis up to Seven Days?
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DTH:19002
Record Dates: First submitted 2019-06-23; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Acute Cholecystitis
Keywords: Acute cholecystitis; Early laparoscopic cholecystectomy; Gallbladder disease; Late laparoscopic cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute; Gallbladder Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E: Early LC (n=60) (Active Comparator): Early laparoscopic cholecystectomy (within 72h from symptom onset)
  Interventions: Procedure: Early laparoscopic cholecystectomy
- Group L: Late LC (n=60) (Active Comparator): Late laparoscopic cholecystectomy (after 72h up to seven days from symptom onset)
  Interventions: Procedure: Late laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Early laparoscopic cholecystectomy — within 72h from symptom onset
  Arms: Group E: Early LC (n=60)
Procedure: Late laparoscopic cholecystectomy — after 72h up to seven days from symptom onset
  Arms: Group L: Late LC (n=60)

SUMMARY:
Objectives: To compare the safety of early (≤72h) versus late (>72h-7days) laparoscopic cholecystectomy (LC) from symptom onset for acute cholecystitis (AC).

Background: As LC within 72h of symptom onset was considered the optimum time, sometimes there was a delay in diagnosis and management. So, we raised the question of safety and feasibility of performing LC to patients with AC who failed to have LC within 72h of acute attack.

Patients and Methods: This was a prospective, randomized, double-blind, clinical trial; carried out on 120 patients presented with AC between September 2017 and April 2019. Patients were randomly allocated into two equal groups assigned to LC; group E: within 72h of symptom onset, and group L: after 72h up to seven days from symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AC within seven days from symptom onset
* American Society of Anesthesiologist (ASA) physical status ≤ II
* Age from 21 to 60 years

Exclusion Criteria:

* Patients with ASA physical status > II
* Age < 21 years or > 60 years
* Child classification B or C
* Choledocholithiasis
* Acute pancreatitis
* Severe sepsis
* Gallbladder perforation
* Pregnant women

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants and Rate of Post-operative complications | 30 days post-operatively
  Number of participants and Rate of: Post-operative bleeding, Fluid collection, Bile leak, Port-site infection, Revision surgery, Mortality rate

SECONDARY OUTCOMES:
Mean and Standard deviation of Operative duration (hours) (mean±SD) | from surgical incision till suture closure
  Mean and Standard deviation of Operative duration (hours)
Mean and Standard deviation of Intra-operative blood loss (ml) (mean±SD) | from surgical incision till suture closure
  Mean and Standard deviation of Intra-operative blood loss (ml)
Number of participants and Rate of Conversion to open cholecystectomy | from the start till the end of surgical procedure
  Number of participants and Rate of Conversion to open cholecystectomy
Mean and Standard deviation of Length of hospital stay (days) (mean±SD) | from hospital admission till home discharge within 30 days
  Mean and Standard deviation of Length of hospital stay (days)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Abdalgaleil, MD, Principal Investigator — Damanhour Teaching Hospital; Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital; Osama S Elbalky, MD, Study Director — Damanhour Teaching Hospital; Mamdouh M Ibrahim, MD, Study Chair — Damanhour Teaching Hospital; Mohamed S Elnagar, MD, Study Chair — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt